CLINICAL TRIAL: NCT06472960
Title: Relationships Between Physical Activity and Inhibitory Control Among College Students: fNIRS and Fundus Imaging
Brief Title: Relationships Between Physical Activity and Inhibitory Control Among College Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen University (Other)
Responsible Party: Principal Investigator, Liye Zou, Professor, Shenzhen University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SZUPaIntervention
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Cognition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate-intensity cycling (Experimental): Moderate-intensity cycling on Ergoline Ergoselect 100
  Interventions: Behavioral: Moderate-intensity cycling; Behavioral: Uninterrupted sitting
- Vigorous-intensity cycling (Experimental): Vigorous-intensity cycling on Ergoline Ergoselect 100
  Interventions: Behavioral: Vigorous-intensity cycling; Behavioral: Uninterrupted sitting
- Uninterrupted sitting (Experimental): Uninterrupted sitting in a quiet room
  Interventions: Behavioral: Uninterrupted sitting

INTERVENTIONS:
Behavioral: Moderate-intensity cycling — Moderate-intensity cycling on Ergoline Ergoselect 100
  Arms: Moderate-intensity cycling
Behavioral: Vigorous-intensity cycling — Vigorous-intensity cycling on Ergoline Ergoselect 100
  Arms: Vigorous-intensity cycling
Behavioral: Uninterrupted sitting — Uninterrupted sitting in a quiet room

SUMMARY:
The primary aim of this study is to explore the impact of a 20-minute aerobic exercise on inhibitory control, microvascular diameters, and brain function. The main questions it aims to answer are:

1. Is there a correlation among the level of physical activity, performance in inhibitory control, and the diameter of retinal microvasculature, and do retinal microcirculation parameters mediate this relationship?
2. Does short-term aerobic exercise (moderate and high intensity) improve inhibitory control and physiological markers, such as retinal diameter and frontal brain activation, compared to a sedentary control group?

ELIGIBILITY:
Inclusion Criteria:

* right-handed (how was handedness assessed; i.e., "What hand do you write with?") with normal or corrected-to-normal vision and normal color vision

Exclusion Criteria:

* reported a history of cardiovascular, metabolic, gastrointestinal, neurological, or psychiatric disorders, medical conditions requiring medical care, substance addiction, strict diets (e.g., low- carbohydrate and Mediterranean diet), pregnancy, or lactation.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | 21 weeks
  This primary outcome measure is assessed by the modified dual-task Stroop paradigm.
Retinal Vessel Diameter | 21 weeks
  Retinal Vessel Diameter is assessed by the fully automated fundus camera.
Brain Connectivity | 21 weeks
  Brain connectivity is assessed by the NIRSport2 device

CONTACTS AND LOCATIONS:
Locations (1):
- Body-Brain-Mind Laboratory, School of Psychology, Shenzhen University, Shenzhen, Guangdong, China